CLINICAL TRIAL: NCT07378293
Title: Effects of Selected Statins on Blood Glucose Levels in Healthy Volunteers: A Randomized Phase I Clinical Trial
Brief Title: Effects of Selected Statins on Blood Glucose Levels in Healthy Volunteers
Acronym: [Statins]
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shaheed Benazir Bhutto University Sheringal Dir Upper (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr Abid Ullah, Lecturer, Shaheed Benazir Bhutto University Sheringal Dir Upper
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBBU/PHM-25-33; SBBU/IREC-25-32 (Other: ShaheedBenazirBhuttoUSheringalDU)
Record Dates: First submitted 2026-01-19; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabete Mellitus; Lipid Profile
MeSH Terms: conditions — Diabetes Mellitus | interventions — Simvastatin; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Intervention Model Description: The drugs Rosuvastatin (5mg, 20mg, 40mg), atorvastatin (10mg,20mg, 40mg) and simvastatin(10mg, 20mg, 40mg) will be given orally to the participants of different assigned groups in once daily dosing for two days to assess the effect on blood glucose.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The PI will give the assigned medication to each participant according to randomization and allocation. All the personnel involved in the study will be kept blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin (5mg, 20mg, 40mg) (Experimental): The assigned participants will be given Rosuvastatin 5mg, 20mg, 40mg OD for two days
  Interventions: Drug: Rosuvastatin (5mg, 20mg, 40mg)
- Atorvastatin (10mg,20mg, 40mg) (Experimental): The assigned participants will be given Atorvastatin 10mg,20mg, 40mg OD for two days
  Interventions: Drug: Atorvastatin (10mg, 20mg, 40mg)
- Simvastatin (10mg, 20mg, 40mg) (Experimental): The assigned participants will be given Simvastatin 10mg, 20mg, 40mg OD for two days
  Interventions: Drug: Simvastatin (10mg, 20mg, 40mg)

INTERVENTIONS:
Drug: Simvastatin (10mg, 20mg, 40mg) — The Simvastatin (10mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Other Names: Simvastatin
  Arms: Simvastatin (10mg, 20mg, 40mg)
Drug: Rosuvastatin (5mg, 20mg, 40mg) — The Rosuvastatin (5mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Other Names: Rosuvastatin
  Arms: Rosuvastatin (5mg, 20mg, 40mg)
Drug: Atorvastatin (10mg, 20mg, 40mg) — The Atorvastatin (10mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Other Names: Atorvastatin
  Arms: Atorvastatin (10mg,20mg, 40mg)

SUMMARY:
This Phase I randomized clinical trial aims to investigate the short-term effects of three commonly prescribed statins (atorvastatin, rosuvastatin, and simvastatin) at different dose levels on blood glucose homeostasis in healthy volunteers. The study will assess changes in fasting blood glucose, insulin, and C-peptide levels following two days of statin administration under controlled conditions. The research seeks to provide comparative data on the potential diabetogenic effects of these medications.

DETAILED DESCRIPTION:
This study addresses emerging evidence suggesting statin therapy may modestly increase diabetes risk in a dose-dependent manner. The trial will enroll healthy volunteers who will be randomized to receive one of three statins at low, moderate, or high doses for two days. Blood glucose will be measured using standardized glucometers, while insulin and C-peptide levels will be determined using ELISA assays. The study aims to clarify whether different statins have varying effects on glucose metabolism during short-term exposure and to establish dose-response relationships.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* Non diabetic
* blood glucose level (less than140 mg/dl)

Exclusion Criteria:

* Participants with a history of diabetes mellitus
* With chronic diseases e.g heart disease, kidney disease
* participants taking other medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Measurements | before dosing and 2 days after dosing
  Blood glucose of the subjects will be determined by glucometer in mg/dl
Insulin Levels Determination | Before dosing and two days after dosing
  Blood insulin levels of each participants will be checked by using human insulin ELISA kit 96 wells on respective peak plasma concentration of respective statin
C- Peptide determination | Before dosing and after two days of Dosing
  Blood samples approx. 4 mL will be taken from the participants to check C- Peptide levels by using human peptide C ELISA kit on respective peak plasma concentration of respective statin

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abid Ullah, PhD, Principal Investigator — Shaheed Benazir Bhutto University,sheringal
Locations (1):
- Shaheed Benazir Bhutto University Sheringal Dir Upper, Dīr, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study results will be shared in Journals without the participant identifiers.
Supporting Information: CSR